CLINICAL TRIAL: NCT04225013
Title: Early Diagnosis as a Strategy in Reducing the Incidence of Acute Renal Failure and Mortality Associated With Contrast Media Administration in Cardiovascular Procedures
Brief Title: Early Diagnosis as Strategy in Reducing the Incidence of Contrast-induced Nephropathy
Status: Completed | Type: Observational
Sponsor: R. Laura Vicente Vicente (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other); Salamanca University Hospital (Other); University of Salamanca (Other)
Responsible Party: Sponsor-Investigator, R. Laura Vicente Vicente, Principal Investigator, Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León
Organization: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Other Study IDs: DIAGNO-CIN
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Kidney Injury; Contrast-induced Nephropathy
Keywords: Biomarker; Contrast-Media; Nephrotoxicity; Prevention; Diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control (no CIN): Patients who receive contrast media but do not develop contrast-induced nephropathy
  Interventions: Diagnostic Test: Early kidney damage biomarkers; Diagnostic Test: Predisposition to kidney injury biomarkers
- Case (yes CIN): Patients who receive contrast media and develop contrast-induced nephropathy
  Interventions: Diagnostic Test: Early kidney damage biomarkers; Diagnostic Test: Predisposition to kidney injury biomarkers

INTERVENTIONS:
Diagnostic Test: Early kidney damage biomarkers — In the urine samples of these patients, a series of biomarkers of early kidney damage and / or predisposition to kidney damage will be measured
  Other Names: N-acetyl-beta-D-glucosaminidase (NAG); Kidney Injury Molecule-1 (KIM-1); Neutrophil gelatinase-associated lipocalin (NGAL); Albumin
Diagnostic Test: Predisposition to kidney injury biomarkers — In the urine samples of these patients, a series of biomarkers of predisposition to kidney damage will be measured

SUMMARY:
Renal damage due to contrast media (CM) administration is one of the main complications of cardiac intervention and is called contrast-induced nephropathy (CIN). Patients suffering from CIN have a high probability of developing acute renal failure. Today there is no treatment capable of reversing kidney damage, so the best strategy is prevention, by early diagnosis. In this regard, a line of research is currently being carried out focused on the identification of new markers capable of detecting susceptibility/predisposition to renal damage before the administration of a potentially nephrotoxic drug, even at doses that alone should not produce Kidney damage. This concept has been called predisposition to kidney damage.

Taking into account all of the above, the objective of this work is to evaluate the ability of the new markers (previously identified in preclinical models) to detect the predisposition to the CIN before administering the CM.

DETAILED DESCRIPTION:
Kidney damage is one of the most frequent complications of cardiac intervention. This pathology is called contrast-induced nephropathy (CIN) and is defined as an increase in plasma creatinine greater than or equal to 0.5 mg/dL, or greater than or equal to 25% with respect to baseline, during the 5 days after contrast medium (CM) administration.

The appearance of acute renal damage significantly increases the health costs associated with interventional procedures. This is derived from the increase in the length of hospital stay, in care units, and from the application of dialysis as the only existing treatment. In the United States, it has been estimated that the development of acute in-hospital renal damage increases health expenditure by $ 7933 per patient per day, mainly due to the increase in hospitalization time. Thus, not only the very early detection, but especially the prevention of acute renal damage are key aspects for the prognosis of the patients, and for the control of the health expenditure associated with them.

Iodized CMs are the leading cause of acute renal damage of toxic origin in humans. CMs produce renal ischemia derived from a vasoconstriction that has two effects: on the one hand reduction of glomerular filtration, and on the other, tubular ischemic damage that amplifies the reduction of filtrate and, with it, renal dysfunction.

Different scales have been proposed to determine the risk of developing CIN, which include different variables such as the presence of arterial hypotension, the use of counterpulsation balloon, the age over 75 years, the presence of anaemia, diabetes, the amount of CM used and renal function. Each item is assigned a certain score in the case of being present in the patient and depending on the final score, the possible risk of contrast nephropathy after the procedure and even the risk of dialysis is estimated. However, these scales are not widely used in clinical practice and their usefulness is doubtful.

Currently the detection of renal damage associated with CM is performed using the plasma creatinine marker. The main drawback of this detection mode is that creatinine levels increase when renal functionality is already altered. In other words, detection occurs when renal functionality has decreased by approximately 70%. This is why new markers capable of detecting damage in their earliest stages are currently being evaluated, when the damage is less widespread. Also in the last decade a new concept of biomarker called a marker of predisposition to kidney damage has emerged. This concept has been revealed after verifying that certain treatments significantly increase the risk of suffering an acute renal failure, and do so in a hidden and silent way.

This susceptibility can be detected by certain markers, which if its usefulness is validated in clinical practice, this assessment would be a very useful tool to classify the risk of patients, individually. Thus the information provided by the predisposition markers would allow a preventive and personalized medicine to be carried out when subjecting patients to a new procedure or treatment potentially harmful to their kidneys.

Taking into account all of the above, the objective of this work is to evaluate the ability of the new predisposition markers (previously identified in preclinical models) to detect patients at risk of suffering CIN before CM administration.

To carry out this purpose, patients who are going to receive an CM will be recruited from the Cardiology Service of the University Assistance Complex of Salamanca (CAUSA). Patients who agree to be part of the study must sign an informed consent.

DATA COLLECTION, SAMPLES AND PROCESSING Each patient is assigned an alphanumeric code, therefore their identity will only be known by the cardiology staff.

At the time of inclusion in the study, the following information will be collected for each patient: date of sample collection, general data, anthropometric data, risk factors, prescribed drugs.

Both before the CM administration and daily for the next 5 days, the plasma creatinine value obtained through the patient's medical history will be collected, since this is a determination that is made as part of the care procedure.

A urine sample will be collected before the CM administration. This sample will be coded with the code mentioned above and will be taken to the CAUSA Sample Bank, where it will be centrifuged, aliquoted and stored at -80 degrees Celsius.

URINE SAMPLES ANALYSIS The following determinations will be made: Proteinuria: marker used in the clinic, the Bradford colorimetric technique will be used; Early kidney damage markers and predisposition markers using colorimetric methods, ELISAs and Western Blot STATISTIC ANALYSIS A significance level of 0.05 will be used. The data analysis will be performed with STATA 10 and Statistical Package for the Social Sciences (SPSS) 23.0. Different contrast will be applied depending on the association that is to be studied in each case, and the type of variables such as: normality test (Kolmogorov-Smirnov, Shapiro-Wilk), frequency comparison (X2), correlation test (Pearson, Spearman), comparison of means for independent data (ANOVA and Kruskal-Wallis) and repeated measures ANOVA and Wilcoxon test for paired data.

STUDY LIMITATIONS Although the study follows all the recommendations for observational studies considered in the STORBE statement (STregthening the Reporting of OBservational studies in Epidemiology), there is a possibility that there are factors that have not been considered. On the other hand, the included variables are biomarkers of early kidney damage and predisposition to acute renal damage induced by certain renal toxins. It is possible that there are other markers (unknown), that there are not being analysed, and that can predict the kidney damage.

CONCLUSION In summary, this project focuses on finding a solution to a problem of high clinical relevance: to diagnose patients at risk of suffering CIN before CM administration. Therefore, it proposes an objective focused on personalized medicine.

This project will be carried out through the generation of a consortium of professionals from different fields, on the one hand researchers, experts in markers of renal damage and on the other, clinicians specialized in the realization of vascular catheterizations.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age who agree to participate in the study an do not comply with any of the exclusion criteria

Exclusion Criteria:

* Patients who are terminally ill
* Patients who do not wish to sign the informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will receive an iodinated contrast medium as part of a diagnostic or interventional procedure
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Urinary N-acetyl-beta-D-glucosaminidase | Time 0: before administration of the contrast media
  It is an enzyme whose urinary excretion is elevated in case of kidney damage. It is capable of detecting damage before the classic plasma creatinine and urea markers. There are no reference values for humans, so the means of patients who do not develop contrast-induced nephropathy (Control group) should be compared with those who develop the damage (Case group)
Urinary Kidney Injury Molecule -1 | Time 0: before administration of the contrast media
  It is a biomarker of early kidney damage. It is able to detect kidney damge in early stages, before the clinical markers creatinine and plasma urea. There are no reference values for humans, so the means of patients who do not develop contrast-induced nephropathy (Control group) should be compared with those who develop the damage (Case group)
Urinary Neutrophil gelatinase-associated lipocalin (NGAL) | Time 0: before administration of the contrast media
  It is a biomarker of early kidney damage. It is able to detect kidney damge in early stages, before the clinical markers creatinine and plasma urea. There are no reference values for humans, so the means of patients who do not develop contrast-induced nephropathy (Control group) should be compared with those who develop the damage (Case group)
Urinary albumin | Time 0: before administration of the contrast media
  It is a biomarker of early kidney damage. It is able to detect kidney damge in early stages, before the clinical markers creatinine and plasma urea. There are no reference values for humans, so the means of patients who do not develop contrast-induced nephropathy (Control group) should be compared with those who develop the damage (Case group)
Urinary biomarkers of predisposition to kidney injury | Time 0: before administration of the contrast media
  It is a group of markers thar are in patent phase so their names can not be mentioned. They are able to detect the susceptibility to kidney damage before administering a nephrotoxic agent. There are no reference values for humans, so the means of patients who do not develop contrast-induced nephropathy (Control group) should be compared with those who develop the damage (Case group)

SECONDARY OUTCOMES:
Contrast-induced nephropathy (CIN) development | Time 0 (baseline, before contrast media) and daily for 5 days after contrast media
  To stratify the patients in each group it is necessary to know whether or not they have developed CIN. The definition of this pathology implies the elevation of the plasma creatinine in 0.5 mg / dl (absolute value) or 20% of the individual baseline value in the 5 days after the contrast media administration.
  Therefore, plasma creatinine will be evaluated both before and 5 days after administration of the contrast media.
Percentage of patients with Risk factor's | These data will be collected once, at time 0 (moment of inclusion in the study)
  The percentage of patients who suffer each of the following pathologies / conditions (risk factors), in each study group, will be consulted through the clinical history: Diabetes mellitus, dyslipidemia, high blood pressure, previous kidney disease, obesity, smoking, alcohol use, drug abuse, drug use
Body weight | These data will be collected once, at time 0 (moment of inclusion in the study)
  Body weight will be measured to each patient and expressed in kilograms
Height | These data will be collected once, at time 0 (moment of inclusion in the study)
  The height will be measured to each patient and expressed in meters
Age | These data will be collected once, at time 0 (moment of inclusion in the study)
  Through the year of birth, the patient's age will be calculated, wich will be expressed in years
Sex | These data will be collected once, at time 0 (moment of inclusion in the study)
  Patients will be classified according sex in Male or Female
Contrast media | These data will be collected once, at day 1 (after contrast media administration)
  The following information regarding the contrast media will be obtained:
  * Name: in each experimental group the percentage of each type of contrast medium will be calculated
  * Volume, in mL: the arithmetic mean of the volumes administered of each type of contrast medium in each experimental group will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Ana Isabel Morales Martín, PhD, Principal Investigator — University of Salamanca
Locations (1):
- Servicio de Cardiología del CAUSA, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vicente-Vicente L, Casanova AG, Hernandez-Sanchez MT, Prieto M, Martinez-Salgado C, Lopez-Hernandez FJ, Cruz-Gonzalez I, Morales AI. Albuminuria Pre-Emptively Identifies Cardiac Patients at Risk of Contrast-Induced Nephropathy. J Clin Med. 2021 Oct 26;10(21):4942. doi: 10.3390/jcm10214942. PMID 34768464